CLINICAL TRIAL: NCT03789916
Title: Single Versus Dual Antiplatelet Therapy in Patients With Incomplete Revascularization After Coronary Artery Bypass Graft Surgery
Brief Title: SAPT Versus DAPT in Incomplete Revascularization After CABG
Acronym: SDAT-IRC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Antonio Nenna, MD, Cardiovascular Surgery, Campus Bio-Medico University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 72.18
Record Dates: First submitted 2018-12-27; First posted 2018-12-31 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery bypass grafting; incomplete revascularization; coronary artery disease; dual antiplatelet therapy
MeSH Terms: conditions — Coronary Artery Disease | interventions — Ticagrelor; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DAPT (Experimental): "Dual antiplatelet therapy": acetylsalicylic acid 100 mg/die + ticagrelor 90 mg bis in die
  Interventions: Drug: Ticagrelor; Drug: acetylsalicylic acid
- SAPT (Active Comparator): "Single antiplatelet therapy": acetylsalicylic acid 100 mg/die
  Interventions: Drug: acetylsalicylic acid

INTERVENTIONS:
Drug: Ticagrelor — 90 mg bis in die
  Other Names: Brilique
  Arms: DAPT
Drug: acetylsalicylic acid — 100 mg die

SUMMARY:
The study aims to compare the efficacy of dual antiplatelet therapy (DAPT) over single antiplatelet therapy (SAPT) in patients with incomplete revascularization after coronary artery bypass graft surgery (CABG).

Before hospital discharge, patients will be 1:1 randomized to SAPT (acetylsalicylic acid 100 mg/die) or DAPT (acetylsalicylic acid 100 mg/die + ticagrelor 90 mg bis in die). DAPT will be continued for 12 months, and ticagrelor will be withdrawn thereafter. Primary endpoint is the evaluation of cardiac-related mortality at 5 years from hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing CABG, ± cardiopulmonary bypass, ± any associated cardiac procedures (valve replacement,...)
* incomplete myocardial revascularization, defined by anatomic or functional criteria
* obtained informed consent

Exclusion Criteria:

* acute coronary syndrome < 12 months from surgery
* dual antiplatelet therapy at hospital admission
* planned procedure to complete myocardial revascularization (e.g. hybrid approach)
* intolerance / unable to take acetylsalicylic acid or ticagrelor
* preoperative atrial fibrillation
* impaired compliance
* planned pregnancy
* history of gastrointestinal bleeding
* chronic kidney disease (eGFR < 30 mL/min/1.73 m2)
* chronic liver disease
* severe heart failure at hospital admission
* active malignancy
* alcohol abuse
* any clinical condition not compatible with the treatment

Exit Criteria:

* postoperative atrial fibrillation requiring anticoagulation
* postoperative hemorrhagic events (stroke, GI bleeding)
* occurrence of contraindications to acetylsalicylic acid or ticagrelor
* surgical treatment requiring DAPT withdrawn
* patient decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2019-01-02 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Cardiac-related mortality | 5 years

SECONDARY OUTCOMES:
Mortality | 5 years
  Overall mortality and non-cardiac-related mortality
Major adverse cardiac and cerebrovascular events (MACCEs) | 5 years
  cardiac-related mortality, myocardial infarction, repeated vessel revascularization, hospitalization for heart failure, major arrhythmias, stroke
Major adverse hemorrhagic events (MAHEs) | 5 years
  stroke, gastrointestinal bleeding, life-threatening bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Chello, MD, Study Chair — Università Campus Bio-Medico di Roma, Rome, Italy
Locations (1):
- Università Campus Bio-Medico di Roma, Rome, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR

REFERENCES:
- [Result] Spadaccio C, Nappi F, Nenna A, Beattie G, Chello M, Sutherland FW. Is it time to change how we think about incomplete coronary revascularization? Int J Cardiol. 2016 Dec 1;224:295-298. doi: 10.1016/j.ijcard.2016.09.055. Epub 2016 Sep 18. PMID 27665400